CLINICAL TRIAL: NCT01468454
Title: A Phase II Safety and Efficacy Study of 18F-L-Fluoro-DOPA PET/CT Scan Localization of Focal Pancreatic Lesions in Children With Hyperinsulinemic Hypoglycemia
Brief Title: Phase II Safety and Efficacy Study of 18FDOPA PET-CT in Children With Hyperinsulinemic Hypoglycemia
Acronym: 18FDOPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Lisa States, Principal Investigator, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-006211
Record Dates: First submitted 2011-10-18; First posted 2011-11-09 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Congenital Hyperinsulinism (CHI); Persistent Hyperinsulinemic Hypoglycemia of Infancy (PHHI)
Keywords: Congenital Hyperinsulinism (CHI); hyperinsulinism; Persistent Hyperinsulinemic Hypoglycemia of Infancy (PHHI); CHI; PHHI; Pancreatectomy; 18F-DOPA; PET/CT scan
MeSH Terms: conditions — Congenital Hyperinsulinism; Hyperinsulinism | interventions — fluorodopa F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- (18F-DOPA) PET/CT imaging (Experimental): Obtain safety and efficacy data on the use of 18-labeled L-fluorodeoxyphenylalanine (18F-DOPA) PET imaging in children with HI for the clinical indication of localizing a focal lesion
  Interventions: Drug: 18 F-DOPA

INTERVENTIONS:
Drug: 18 F-DOPA — 1 time injection of 0.08 - 0.16 mCi/kg of 18F-DOPA
  Other Names: 18FDOPA PET SCAN

SUMMARY:
Children with congenital hyperinsulinism (CHI) have low blood sugar, and some of these children may require surgery to remove part or all of their pancreas. In this study, researchers will test how well a radioactive drug, 18-labeled L-fluorodeoxyphenylalanine (called F-DOPA) can detect a form of hyperinsulinism (focal HI) that may be cured by surgery. Eligible participants in this study will have positron emission tomography/computerized tomography (PET/CT) scans with F-DOPA prior to surgery.

DETAILED DESCRIPTION:
For children with congenital hyperinsulinism (CHI), low blood sugar is caused by cells in the pancreas that release too much insulin. Some children with CHI have these cells throughout their pancreas (called diffuse disease); others have them located in specific areas of the pancreas (called focal disease). Children who have focal disease located in specific areas of the pancreas may be cured with surgery. F-DOPA is a radioactive drug that is picked up by these cells and used for positron emission tomography (or PET), an imaging technique used in nuclear medicine departments. In this study, researchers will validate the efficacy and safety of using PET/CT with F-DOPA in the pre-operative localization of focal disease in children with hyperinsulinism.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children with a clinical diagnosis of hyperinsulinism who are suspected to have focal disease and are surgical candidates for pancreatectomy

Exclusion Criteria:

* Pregnant or lactating females
* Any other major illness or condition that might substantially increase the risk associated with the subject's participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-01; Primary Completion 2014-06 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J States, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Hardy OT, Hernandez-Pampaloni M, Saffer JR, Suchi M, Ruchelli E, Zhuang H, Ganguly A, Freifelder R, Adzick NS, Alavi A, Stanley CA. Diagnosis and localization of focal congenital hyperinsulinism by 18F-fluorodopa PET scan. J Pediatr. 2007 Feb;150(2):140-5. doi: 10.1016/j.jpeds.2006.08.028. PMID 17236890
- [Background] Hardy OT, Hernandez-Pampaloni M, Saffer JR, Scheuermann JS, Ernst LM, Freifelder R, Zhuang H, MacMullen C, Becker S, Adzick NS, Divgi C, Alavi A, Stanley CA. Accuracy of [18F]fluorodopa positron emission tomography for diagnosing and localizing focal congenital hyperinsulinism. J Clin Endocrinol Metab. 2007 Dec;92(12):4706-11. doi: 10.1210/jc.2007-1637. Epub 2007 Sep 25. PMID 17895314
- [Background] Hardy OT, Litman RS. Congenital hyperinsulinism - a review of the disorder and a discussion of the anesthesia management. Paediatr Anaesth. 2007 Jul;17(7):616-21. doi: 10.1111/j.1460-9592.2007.02192.x. PMID 17564642
- [Background] Peranteau WH, Ganguly A, Steinmuller L, Thornton P, Johnson MP, Howell LJ, Stanley CA, Adzick NS. Prenatal diagnosis and postnatal management of diffuse congenital hyperinsulinism: a case report. Fetal Diagn Ther. 2006;21(6):515-8. doi: 10.1159/000095664. Epub 2006 Sep 12. PMID 16969006
- [Background] Chevalme, Yanna-Marina et al. FDOPA-(18F): a PET radiopharmaceutical recently registered for diagnostic use in countries of the European Union. Braz. arch. biol. technol. [online]. 2007, vol.50, n.spe [cited 2011-10-06], pp. 77-90 . Available from: <http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1516-89132007000600009&lng=en&nrm=iso>. ISSN 1516-8913. http://dx.doi.org/10.1590/S1516-89132007000600009.
- [Result] Laje P, States LJ, Zhuang H, Becker SA, Palladino AA, Stanley CA, Adzick NS. Accuracy of PET/CT Scan in the diagnosis of the focal form of congenital hyperinsulinism. J Pediatr Surg. 2013 Feb;48(2):388-93. doi: 10.1016/j.jpedsurg.2012.11.025. PMID 23414871
- [Result] Laje P, Palladino AA, Bhatti TR, States LJ, Stanley CA, Adzick NS. Pancreatic surgery in infants with Beckwith-Wiedemann syndrome and hyperinsulinism. J Pediatr Surg. 2013 Dec;48(12):2511-6. doi: 10.1016/j.jpedsurg.2013.05.016. PMID 24314195
- [Result] Peranteau WH, Palladino AA, Bhatti TR, Becker SA, States LJ, Stanley CA, Adzick NS. The surgical management of insulinomas in children. J Pediatr Surg. 2013 Dec;48(12):2517-24. doi: 10.1016/j.jpedsurg.2013.04.022. PMID 24314196
- See also: The Congenital Hyperinsulinism Center at The Children's Hospital of Philadelphia — http://www.chop.edu/service/congenital-hyperinsulinism-center/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2009 to July 2013, the study team recruited and enrolled 129 subjects referred to the Congenital Hyperinsulinism Center at the Children's Hospital of Philadelphia who were potential candidates for partial pancreatectomy surgery if focal lesions were suspected and were able to be localized.
Pre-assignment Details: 1 subject was enrolled into the study (informed consent signed), however, was deemed ineligible due to subsequent additional clinical information provided after consent but prior to scheduled PET study. . A second subject had two scans, but is only counted once in the final analysis. This accounts for the enrollment discrepancy (130 vs.128 described in the protocol section)
Groups:
- F-DOPA PET/CT Imaging vs Surgical Result: 18 F-DOPA: 1 time injection of 0.08 - 0.16 mCi/kg of 18F-DOPA given 10-15 minutes prior image acquisition.
Period: Overall Study
Arm/Group | F-DOPA PET/CT Imaging vs Surgical Result
Started | 128
PETs Completed | 128
Had Both PET and Surgery | 119
Completed | 119
Not Completed | 9
Not completed — Did not have surgery after PET | 9

BASELINE CHARACTERISTICS:
Population: Subjects referred to the Congenital Hyperinsulinism Center at the Children's Hospital of Philadelphia from January 2009 to July 2013 for evaluation, diagnosis, treatment and potential surgery for Congenital HI
Groups:
- (18F-DOPA) PET/CT Imaging vs Surgical Results: 18 F-DOPA: 1 time injection of 0.08 - 0.16 mCi/kg of 18F-DOPA given 10-15 minutes prior image acquisition.
Arm/Group | (18F-DOPA) PET/CT Imaging vs Surgical Results
Number analyzed (Participants) | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 128
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 95
  More than one race | 12
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 121
  Canada | 4
  Australia | 1
  Israel | 1
  Paraguay | 1

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of 18F-DOPA PET/CT Scans to Detect Focal Lesions in Children With Congenital Hyperinsulinism
Description: To determine the sensitivity and specificity of 18F-DOPA PET/CT for the detection of a focal pancreatic lesion in infants and children with poorly controlled hyperinsulinemic hypoglycemia.
Time Frame: Surgery typically occured within a week post PET
Population: A single F-DOPA PET/CT imaging study was performed and reported prior to surgery. This data includes surgical histopathology confirmed as focal or diffuse. 19 of the 119 participants with surgical results had atypical histopathology that did not fit the definition of either category and therefore are excluded from this analysis.
Measure: Number; unit: cases
Groups:
- PET/CT Imaging vs Surgical Result: PET/CT imaging results in patients with surgical histologic confirmation.
Arm/Group | PET/CT Imaging vs Surgical Result
Number analyzed (Participants) | 100
cases
  True Negatives (PET diffuse/surgery diffuse) | 34
  False negatives (PET diffuse/surgery focal): | 10
  False positives (PET focal/surgery diffuse): | 4
  True positives (PET focal/surgery focal): | 52
Statistical Analysis 1: Comparison: PET/CT Imaging vs Surgical Result; Test type: Other; Specificity = 89.5, 95% CI 2-sided [75.2 to 97.1]
Statistical Analysis 2: Comparison: PET/CT Imaging vs Surgical Result; Test type: Other; Sensitivity = 83.9, 95% CI 2-sided [72.3 to 92]

2. Secondary Outcome: Safety of 18F-DOPA PET/CT Scan - Number of Participants With Adverse Events
Description: To further evaluate the safety of 18-labeled L-fluorodeoxyphenylalanine (18F-DOPA) PET/CT imaging in infants and children with congenital hyperinsulinism
  - subjects are monitored clinically for any signs or symptoms of adverse events for 72 hours post PET. Adverse events are documented and followed to resolution
Time Frame: evaluated with 72 hours or prior to pancreatic surgery (if any)
Population: all participants who had both PET and surgery
Measure: Count of Participants; unit: Participants
Arm/Group | (18F-DOPA) PET/CT Imaging
Number analyzed (Participants) | 119
Participants | 0

ADVERSE EVENTS:
Time Frame: reviewed within 72 hours post PET or prior to pancreatic surgery (which ever was first)
Description: included all participants who had PET (whether or not they also had surgery)
Arm/Group | (18F-DOPA) PET/CT Imaging
All-Cause Mortality (participants affected / at risk) | 0/128
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes